CLINICAL TRIAL: NCT01722695
Title: HD Performance Comparison of Revaclear 200 and Revaclear 400 With Larger-surface Competitor Dialyzers
Brief Title: Performance Comparison of Revaclear With Larger Dialyzer
Acronym: Revacom HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1499
Record Dates: First submitted 2012-10-22; First posted 2012-11-07 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Revaclear followed by FX (Other)
  Interventions: Other: Dialyzer comparison
- FX followed by Revaclear (Other)
  Interventions: Other: Dialyzer comparison

INTERVENTIONS:
Other: Dialyzer comparison — Each patient is treated by hemodialysis for one week (3 sessions) with each dialyzer type (Revaclear or FX).
  The order of dialyzers used will be randomly assigned to the patient at randomization.

SUMMARY:
The purpose of the study is to show equivalent performance of the Revaclear dialyzer when compared to a dialyzer with larger membrane surface area.

Study design: open, randomized, cross-over, multicentric, controlled prospective

Medical devices: Revaclear 200 versus FX 60 or Revaclear 400 versus FX 100, depending on patient needs

Patients/sample size: 30 adult chronic hemodialysis patients

Treatment: Each patient will be treated by hemodialysis for one week (3 dialysis sessions) with Revaclear dialyzers and one week (3 dialysis sessions) with FX dialyzers.

Objectives: intraindividual comparison of dialysis dose; reduction rates and total removal of urea, phosphate, creatinine and ß2-microglobulin; albumin loss

Primary variable: dialysis dose Kt/V urea

Secondary variable: reduction rates and total removal of urea, phosphate, creatinine and ß2-microglobulin

Safety variable: albumin loss, blood count

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure and stable treatment with hemodialysis or hemodiafiltration for at least 3 months
* patients aged 18 years or more
* written consent to participate in the study (informed consent)
* dialysis via native fistula or Gore-Tex graft capable of providing a blood flow rate of at least 300 mL/min

Exclusion Criteria:

* single-needle dialysis
* pregnant and lactating women
* participation in other interventional studies less than 3 months prior to study start
* non-compliance with the dialysis prescription
* hematocrit less than 28%
* hospitalization
* antibiotic therapy
* active infection
* active cancer
* known positive serology for HIV, hepatitis B or C
* serious hemostasis disorders
* any comorbidity possibly conflicting with the study purpose or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Dialysis dose Kt/V urea | 2 weeks (6 consecutive dialysis sessions)
  Calculation from pre and post plasma urea concentration or urea nitrogen, session length, ultrafiltration volume and post dialysis weight. Dialysis dose does not have a unit of measure.

SECONDARY OUTCOMES:
Reduction rate of urea, creatinine, phosphate and ß2-microglobulin | 2 weeks (6 consecutive dialysis sessions)
  Calculation from pre and post dialysis plasma concentrations. Unit of measure is percentage (%).
Total removal of creatinine, phosphate and ß2-microglobulin | 2 weeks (6 consecutive dialysis sessions)
  Calculation from measured concentration in integrated dialysate sample over entire treatment, dialysate flow rate, treatment duration and ultrafiltration volume. Unit of measure is g or mg per treatment.
Albumin loss | 2 weeks (6 consecutive dialysis sessions)
  Calculation from measured concentration in integrated dialysate sample over entire treatment, dialysate flow rate, treatment duration and ultrafiltration volume. Unit of measure is g or mg per treatment.

OTHER OUTCOMES:
Blood count | 2 weeks (start and end of 6 consecutive dialysis sessions)
  Parameters are hemoglobin concentration (g/dL), hematocrit (%), thrombocyte concentration (G/L), erythrocyte concentration (T/L), leukocyte concentration (G/L).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rosenkranz, Prof., Principal Investigator — Medical University Graz, Austria
Locations (2):
- Austria (2):
  - Dialyseinstitut Prim. Dr. W. Gießauf GmbH, Graz
  - Medical University Graz, Graz